CLINICAL TRIAL: NCT05614414
Title: Postoperative Sore Throat: Interest of the Videolaryngoscope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mongi Slim Hospital (Other)
Responsible Party: Principal Investigator, Mhamed Sami Mebazaa, Professor, Mongi Slim Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Sore throat videolaryngoscope
Record Dates: First submitted 2022-10-07; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Sore-throat; Anesthesia; Postoperative Pain; Tracheal Intubation Morbidity
MeSH Terms: conditions — Pharyngitis; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VL Group (Experimental): Patients who were intubated by videolaryngoscope.
  Interventions: Procedure: tracheal intubation by Videolaryngoscope
- LD Group (Active Comparator): Patients who were intubated by direct laryngoscope
  Interventions: Procedure: tracheal intubation by direct laryngoscope

INTERVENTIONS:
Procedure: tracheal intubation by Videolaryngoscope — The investigators performed laryngoscopy using a McGrath video-laryngoscope with a number 4 blade.
  Arms: VL Group
Procedure: tracheal intubation by direct laryngoscope — The investigators performed laryngoscopy using either a Macintosh laryngoscope using a number 4 blade.
  Arms: LD Group

SUMMARY:
Postoperative sore throat is a complication of orotracheal intubation. The aim of our study was to assess the impact of videolaryngoscopy on postoperative sore throat during the first 24 hours following surgery.

This was a prospective, randomized study, over a period of 9 months. The investigators included 136 patients with non-difficult airway, classified ASA I to III and over 18 years old. The patients were randomized into 2 groups: the VL group including 70 patients intubated with direct laryngoscopy and the LD group including 66 patients intubated with videolaryngoscopy.

DETAILED DESCRIPTION:
The investigators monitored blood pressure, ECG, saturation in oxygen, capnograph, temperature and curarization. They also monitored cuff pressure using manometer.

The investigators pre-oxygenated the patients until the fractional expired oxygen was over 90%, then induced anaesthesia using either 2.5 to 3.5 mg/kg of propofol or 0.3 to 0.4 mg/kg of etomidate, then 1mg/kg of suxamethonium (in absence of contraindication). If modified crash induction was performed, the anaesthesiologist mentioned the opioid used.

The investigators performed laryngoscopy using either a Macintosh laryngoscope using a number 4 blade in LD group, or a McGrath video-laryngoscope with a number 4 blade in VL group and a stylet when needed. Women were intubated using number 7 tube and man using a 7.5 tube. They inflated the cuff with 7ml of air, and controlled pressure by manometer every 30 minutes in order to maintain it between 20 and 25 mmHg.

The investigators ventilated patients with assisted controlled mode using a 6ml/kg of ideal weight volume, a 6 mmHg PEEP, a 50% inspired fraction of oxygen and a respiratory rate guaranteeing an end-expiratory CO2 level between 35 and 40 mmHg. Then, they administrated 4 mg of Ondansetran in order to prevent postoperative nausea and vomiting (PONV).

The investigators maintained anaesthesia using either isoflurane or sevoflurane, 0.1 μg/kg of sufentanil and 0.05 mg/kg of atracurium.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years old;
* Patients with ASA status 1, 2 or 3;
* Patients who underwent surgery with general anaesthesia and intubation;
* written consent.

Exclusion Criteria:

* Patients under corticosteroids;
* Pregnant women;
* Patient with at least two difficult intubation criteria or a limited mouth opening (under 2cm), difficult airway management history, upper airway tumour or cervical rachis trauma;
* Patients who had an otorhinolaryngologic infection in the last month, an intubation or endoscopy of upper airway in the last 48 hours, vomiting in the last 24 hours, a gastric tube in the last 24 hours or throat symptoms prior to surgery;
* Patients scheduled for a surgery implying a manipulation of upper airways;
* Patient scheduled for a surgery > 2 hours.

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Postoperative sore throat | 6 hours after surgery
  Postoperative sore throat assessed by verbal scale (from 0 to 10)

SECONDARY OUTCOMES:
Postoperative sore throat | up to 24 hours after surgery.
  Postoperative sore throat assessed by verbal scale (from 0 to 10)
Postoperative dysphonia | up to 24 hours after surgery
  Presence or no of dysphonia
Postoperative dysphagia | up to 24 hours after surgery
  presence or no of dysphagia

CONTACTS AND LOCATIONS:
Locations (1):
- Mongi Slim University Hospital, La Marsa, Tunis Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: No